CLINICAL TRIAL: NCT03149445
Title: A Double-Blind, Randomized, Placebo-Controlled, Multiple-Dose, Multi-Center Safety and Efficacy Study of Co-Administration of Tesofensine/Metoprolol for 12 Weeks in Adult and Adolescent Patients With Prader-Willi Syndrome (PWS), Followed by Two Open Label 12 Weeks Extension Periods for Adolescent Patients
Brief Title: Co-administration of Tesofensine/Metoprolol in Subjects With Prader-Willi Syndrome (PWS)
Acronym: 2016-003694-18
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TM002
Record Dates: First submitted 2017-04-03; First posted 2017-05-11 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Confirmed Genetic Diagnosis of Prader-Willi Syndrome
MeSH Terms: interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Intervention Model Description: Two-centre, double-blind, placebo-controlled, randomized, and multiple-dose clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tesofensine/Metoprolol (Experimental): Tesofensine + metoprolol administered once a day, in the morning with a meal
  Interventions: Drug: Tesofensine/Metoprolol
- Tesofensine/Metoprolol placebo (Placebo Comparator): Placebo tablets matching tesofensine + metoprolol administered once a day, in the morning with meal
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tesofensine/Metoprolol — Study medication will be administered for 91 days.
  Other Names: Tesofensine; Metoprolol
  Arms: Tesofensine/Metoprolol
Drug: Placebos — Study medication will be administered for 91 days.
  Other Names: Placebo
  Arms: Tesofensine/Metoprolol placebo

SUMMARY:
Two-centre, double-blind, placebo-controlled, randomized, and multiple-dose clinical study followed by two open label extension periods.

DETAILED DESCRIPTION:
Two-centre, double-blind, placebo-controlled, randomized, and multiple-dose clinical study. Study medication will be administered for 91 days. The study will be conducted in two steps:

* Step 1 - 9 adult subjects with PWS was treated.
* Sponsor review - following the completion of the treatment of the adult subjects, unblinded efficacy, safety, Pharmacokinetic (PK) data as well as all data from the study in subjects with type 2 diabetes (TM001) will be reviewed by sponsor and an interim analysis will be done. Following competent authority positive opinion regarding the interim analysis and unblinded data the study will proceed to:
* Step 2 - 9 adolescent subjects with PWS was treated.
* OLE (Open Label Extension) I - Participation in a 12-week OLE I was offered to subjects who completed Step 2. 8 subjects entered OLE I.
* OLE (Open Label Extension) II - Participation in a 12-week OLE II was offered to subjects who completed OLE I. 6 subjects continued to OLE II.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with a confirmed genetic diagnosis of Prader-Willi syndrome
2. Age:

   1. Step 1: Adults aged 18-30
   2. Step 2: Adolescents aged 12-17
3. Body Mass Index (BMI):

   1. Step 1: Adults with ≥25 kg/m2
   2. Step 2: Children with a BMI >85th percentile for the same age and sex
4. Normal Blood Pressure (BP) or well managed hypertension (only if dose of BP medication(s) has been stable for >2 months)
5. Normal lipid profile or well managed dyslipidemia (only if dose of lipid-lowering medication(s) has been stable for >2 months)
6. Growth hormone is allowed; but patient must be on stable dose of growth hormone >2 months
7. Type 2 diabetes is allowed, but the following criteria must be met:

   1. HbA1c <10.0 % not being managed with insulin within the past 3 months
   2. Patients taking GLP-1 analogues (e.g. exenatide, liraglutide) must have been on stable dose for >3 months
   3. Fasting plasma glucose <11.0 mmol/l

Exclusion Criteria:

1. BP:

   1. Step 1: Adults with >140/90
   2. Step 2: Adolescents with ≥95th percentile for gender, age, and height
2. Heart Rate (HR) ≥ 90, <50 bpm
3. Hypersensitivity to tesofensine/metoprolol
4. Type 1 diabetes
5. Heart failure New York Heart Association (NYHA) level II or greater, decompensated heart failure
6. Previous myocardial infarction or stroke
7. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other DSM-III disorders, or any other psychiatric condition, which in the investigator's opinion will interfere significantly with study compliance
8. History of major depressive disorder or suicidality
9. Any clinically significant cardiac arrhythmia
10. Treatment with calcium channel blockers and beta blockers
11. Concomitant use of monoaminooxidase inhibitors
12. Bulimia or anorexia nervosa
13. Any agent used for weight loss in the past 3 months
14. Untreated hypo- or hyperthyroidism
15. Clinically significant liver (>3x ULN (Upper Limit of Normal range)) and/or kidney impairment
16. More than 5% weight loss within the last 3 months
17. Any other clinically meaningful condition, in the opinion of the investigator, which would make participation potentially unsafe
18. Contraindications to administration of metoprolol per current Summary of Product Characteristics

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, MD, DMSc, Study Director — Saniona
Locations (2):
- Motol University Hospital, Prague, Czechia
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tesomet 0.50/50 mg: Subjects (adults) were randomized to receive co-administration of 0.5 mg tesofensine/50 mg metoprolol (active medication Tesomet) once daily for 91 days (+2 days after the final assessments with halfdose of metoprolol) during Step 1.
- Placebo (Adult): Subjects (adults) were randomized to receive placebo once daily for 91 days during Step 1.
- Tesomet 0.125/25 mg (DB): Subjects (adolescents) were randomized to receive co-administration of 0.125 mg tesofensine/25 mg metoprolol (active medication Tesomet) once daily for 91 days: +2days after the final assessments with halfdose.
- Placebo (Adolescent): Subjects (adolescents) were randomized to receive placebo once daily for 91 days.
- Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg; Placebo -> Tesomet 0.125/25 mg: Participation in a 12-week OLE I was offered to patients who completed Step 2. Patients were receiving co-administration of 0.125 mg tesofensine/25 mg metoprolol (active medication Tesomet) once daily for 12 weeks during OLE I.
- Tesomet 0.25/25 mg: Participation in a 12 week OLE II was offered to all eligible patients of OLE I. Patients were receiving co-administration of 0.25 mg tesofensine/25 mg metoprolol (active medication Tesomet) once daily for 12 weeks during OLE II.
- Tesomet 0.125/25 mg (OLE II): Participation in a 12 week OLE II was offered to all eligible patients of OLE I. Patients were receiving co-administration of 0.125 mg tesofensine/25 mg metoprolol (active medication) once daily for 12 weeks.
Period: Double-blind (DB) Step 1
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Started | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind (DB) Step 2
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Started | 0 | 0 | 5 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 5 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Extension (OLE) I
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Started | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Open Label Extension (OLE) II
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Total
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants] — Population: It is the same adolescent subjects participating in DB Step 2, OLE I and OLE II.
  Participants
    <=18 years | 0 | 0 | 5 | 4 | 9
    Between 18 and 65 years | 6 | 3 | 0 | 0 | 9
    >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 2 | 10
  Male | 2 | 1 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 3 | 5 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 2 | 3 | 2 | 10
  Czechia | 3 | 1 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to End of Treatment in Mean Body Weight
Description: Percent change from baseline to end of treatment in mean body weight. LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: 5 patients started on Tesomet 0.25/25mg in OLE II however 1 subject discontinued early without any further observations and data are therefore only available from 4 subjects.
Measure: Mean (Standard Deviation); unit: Percent (%) change in mean body weight
Groups:
- Tesomet 0.25/25 mg: Participation in a 12 week OLE II was offered to all eligible patients of OLE I. Patients were receiving coadministration of 0.25 mg tesofensine/25 mg metoprolol (active medication Tesomet) once daily for 12 weeks during OLE II.
- Tesomet 0.125/25 mg (OLE II): Participation in a 12 week OLE II was offered to all eligible patients of OLE I. Patients were receiving coadministration of 0.125 mg tesofensine/25 mg metoprolol (active medication) once daily for 12 weeks.
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 4 | 1
Percent (%) change in mean body weight | -4.09 (3.73) | -0.38 (2.05) | 3.56 (2.73) | 3.00 (2.35) | 5.79 (2.08) | 0.33 (3.26) | -1.20 (3.80) | -5.51 (NA) — Only 1 subject was included in this group.
Statistical Analysis 1: Comparison: Tesomet 0.50/50 mg vs Placebo (Adult); Test type: Superiority; p = 0.1045, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = -5.4, 95% CI 2-sided [-12.3 to 1.5]
Statistical Analysis 2: Comparison: Tesomet 0.125/25 mg (DB) vs Placebo (Adolescent); Test type: Superiority; p = 0.7422, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 0.7, 95% CI 2-sided [-4.0 to 5.3]
Statistical Analysis 3: Comparison: Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg vs Placebo -> Tesomet 0.125/25 mg; Test type: Superiority; p = 0.0460, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 5.6, 95% CI 2-sided [0.1 to 11.0]
Statistical Analysis 4: Comparison: Tesomet 0.25/25 mg vs Tesomet 0.125/25 mg (OLE II); Test type: Superiority; p = 0.3847, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 4.3, 95% CI 2-sided [-9.2 to 17.8]

2. Secondary Outcome: Change From Baseline to End of Treatment in Mean Body Weight
Description: Change from baseline to end of treatment in body weight [kg]. LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 4 | 1
kg | -4.15 (4.82) | -0.77 (3.23) | 3.10 (2.85) | 2.25 (1.71) | 4.75 (2.41) | 0.45 (2.82) | -0.90 (3.20) | -3.50 (NA) — Only 1 subject was included in this group.
Statistical Analysis 1: Comparison: Tesomet 0.50/50 mg vs Placebo (Adult); Test type: Superiority; p = 0.1326, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = -6.2, 95% CI 2-sided [-14.9 to 2.5]
Statistical Analysis 2: Comparison: Tesomet 0.125/25 mg (DB) vs Placebo (Adolescent); Test type: Superiority; p = 0.5148, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 1.2, 95% CI 2-sided [-2.9 to 5.3]
Statistical Analysis 3: Comparison: Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg vs Placebo -> Tesomet 0.125/25 mg; Test type: Superiority; p = 0.0605, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 4.5, 95% CI 2-sided [-0.3 to 9.4]
Statistical Analysis 4: Comparison: Tesomet 0.25/25 mg vs Tesomet 0.125/25 mg (OLE II); Test type: Superiority; p = 0.5198, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 2.6, 95% CI 2-sided [-8.8 to 14.0]

3. Secondary Outcome: Change From Baseline to End of Treatment in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) Score
Description: Change from baseline to end of treatment in HQ-CT score. LOCF. HQ-CT score was based upon a questionnaire with 9 items, each of them yielding a score between 0 and 4 resulting in a maximum HQ-CT score of 36. Change in HQ-CT answers (by question and in total) calculated as score at visit 2, 5, 9 or 14 minus score at screening visit 1 was analysed and presented using standard descriptive statistics (mean, median, standard deviation, minimum and maximum value). A decrease in total score indicates an improvement in hyperphagia. If less than three questions were answered by a subject, the missing answers were imputed by the mean score of all other available answers. In case of more than three missing answers, the total score was not calculated. For further information please refer to protocol appendix section 17.1.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: Data only available for 2 patients in Step I placebo arm. 5 patients started on Tesomet 0.25/25mg in OLE II however 1 subject discontinued early without any further observations and data are therefore only available from 4 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 2 | 5 | 4 | 4 | 4 | 4 | 1
score on a scale | -8.50 (9.25) | -4.00 (7.07) | -3.30 (6.82) | -6.75 (3.69) | 1.25 (5.68) | -1.75 (1.50) | -1.00 (2.00) | -2.00 (NA) — Only 1 subject was included in this group.
Statistical Analysis 1: Comparison: Tesomet 0.50/50 mg vs Placebo (Adult); Test type: Superiority; p = 0.0058, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = -8.1, 95% CI 2-sided [-12.5 to -3.6]
Statistical Analysis 2: Comparison: Tesomet 0.125/25 mg (DB) vs Placebo (Adolescent); Test type: Superiority; p = 0.5142, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 2.1, 95% CI 2-sided [-5.3 to 9.5]
Statistical Analysis 3: Comparison: Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg vs Placebo -> Tesomet 0.125/25 mg; Test type: Superiority; p = 0.3794, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 3.1, 95% CI 2-sided [-5.1 to 11.3]
Statistical Analysis 4: Comparison: Tesomet 0.25/25 mg vs Tesomet 0.125/25 mg (OLE II); Test type: Superiority; p = 0.6850, ANCOVA — P-value from an ANCOVA with treatment as factor and baseline as covariate; LS Mean Difference = 1.0, 95% CI 2-sided [-6.1 to 8.1]

4. Secondary Outcome: Steady State Concentrations of Tesofensine and Metoprolol as Measured by Trough Values
Description: Steady state concentrations of tesofensine and metoprolol as measured by trough values. Observed values.
Time Frame: DB Step 1: Day 29; DB Step 2: Day 29; OLE I: Day 120; OLE II: Day 210
Population: No data available for placebo arm in Step I and Step 2. Data only available for 3 patients in OLE I (Placebo -> Tesomet 0.125/25 mg). 5 patients started on Tesomet 0.25/25mg in OLE II however 1 subject discontinued early without any further observations and data are therefore only available from 4 subjects.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 0 | 5 | 0 | 4 | 3 | 4 | 1
μg/L
  Tesofensine | 16.29 (49.8) |  | 3.34 (32.2) |  | 4.14 (17.3) | 5.06 (18.0) | 4.13 (137.5) | 6.43 (NA) — Only 1 subject was included in this group.
  Teso. metab. | 2.97 (52.6) |  | 0.79 (17.1) |  | 1.45 (23.3) | 1.00 (41.9) | 1.56 (49.1) | 1.98 (NA) — Only 1 subject was included in this group.
  Metoprolol | 1.61 (903.7) |  | 1.97 (285.5) |  | 2.81 (119.0) | 3.32 (32.0) | 1.76 (242.5) | 14.50 (NA) — Only 1 subject was included in this group.

5. Secondary Outcome: Change From Baseline to End of Treatment in Fat- and Fat Free Mass (%) by Dual X-ray Absorptiometry (DEXA)
Description: Change from baseline to end of treatment in fat- and fat free mass (%) by dual X-ray absorptiometry (DEXA). Observed values.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: Data only available for 3 patients in Step I (Tesomet 0.50/50 mg). Data not available for the Placebo (adult) arm. Data only available for 3 patients in Step 2 (Tesomet 0.125/25 mg (DB)). Data only available for 2 patients in Step 2 (Placebo (adolescent)). Data only available for 3 patients in OLE I (Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg).
  Data only available for 2 patients in OLE I (Placebo -> Tesomet 0.125/25 mg). Data only available for 2 patients in OLE II (Tesomet 0.25/25 mg).
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 3 | 0 | 3 | 2 | 3 | 2 | 2 | 1
Percent (%)
  Fat mass | -1.27 (1.07) |  | -0.13 (0.25) | -0.50 (0.85) | 1.20 (1.74) | -0.05 (0.21) | -1.70 (0.1) | -1.50 (NA) — Only 1 subject was included in this group.
  Fat free mass | 1.19 (1.11) |  | 0.137 (0.217) | -2.080 (4.511) | 0.053 (2.559) | 4.290 (3.974) | 0.000 (0.1) | 1.470 (NA) — Only 1 subject was included in this group.

6. Secondary Outcome: Change From Baseline to End of Treatment in Bone Mineral Density (BMD) by Dual X-ray Absorptiometry (DEXA)
Description: Change from baseline to end of treatment in BMD by dual X-ray absorptiometry (DEXA). Observed values.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 3 | 0 | 3 | 2 | 3 | 2 | 2 | 1
g/cm^2 | 0.002 (0.0017) |  | 0.019 (0.009) | 0.035 (0.008) | -0.006 (0.008) | -0.007 (0.009) | 0.023 (0.0) | 0.009 (NA) — Only 1 subject was included in this group.

7. Secondary Outcome: Change From Baseline to End of Treatment in Bone Mineral Content (BMC) by Dual X-ray Absorptiometry (DEXA)
Description: Change from baseline to end of treatment in BMC by dual X-ray absorptiometry (DEXA). Observed values.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 3 | 0 | 3 | 2 | 3 | 2 | 2 | 1
gram | 9.5 (63.8) |  | 74.77 (22.46) | 35.53 (55.37) | -1.12 (17.86) | 5.69 (66.33) | 22.51 (46.6) | -21.90 (NA) — Only 1 subject was included in this group.

8. Secondary Outcome: Change From Baseline to End of Treatment in Heart Rate (HR)
Description: Change from baseline to end of treatment in HR (bpm). LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 4 | 1
bpm | 8.22 (4.26) | 7.89 (7.88) | 5.87 (11.01) | 2.75 (8.96) | 2.42 (15.14) | 0.33 (8.65) | -9.50 (10.86) | -5.67 (NA) — Only 1 subject was included in this group.

9. Secondary Outcome: Change From Baseline to End of Treatment in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline to end of treatment in SBP (mmHg) and DBP (mmHg). LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 4 | 1
mmHg
  Change in SBP | -2.72 (9.96) | 0.11 (15.22) | -0.13 (15.79) | -5.00 (9.26) | 5.67 (11.30) | 8.08 (6.45) | -5.33 (2.60) | -9.67 (NA) — Only 1 subject was included in this group.
  Change in DBP | 0.94 (10.72) | -8.89 (8.00) | -1.07 (7.06) | 0.33 (2.54) | 2.92 (10.22) | 4.00 (5.40) | -6.42 (3.95) | 1.33 (NA) — Only 1 subject was included in this group.

10. Secondary Outcome: Total Number of Adverse Events
Description: Total number of Adverse Events
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Measure: Number; unit: Total number of adverse events
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 5 | 1
Total number of adverse events | 23 | 10 | 19 | 9 | 11 | 12 | 14 | 5

11. Secondary Outcome: Change From Baseline to End of Treatment in PR Interval
Description: Change from baseline to end of treatment in PR interval. Observed values.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: Data only available for 1 patient in Step I (Tesomet 0.50/50 mg). Data not available for the Placebo (adult) arm. Data only available for 1 patient in Step 2 (Tesomet 0.125/25 mg (DB)). Data only available for 2 patients in Step 2 (Placebo (adolescent)). Data only available for 1 patient in OLE I (Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg).
  Data only available for 1 patient in OLE I (Placebo -> Tesomet 0.125/25 mg). Data not available for OLE II (Tesomet 0.25/25 mg).
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1
ms | -20.0 (NA) — Only 1 subject was included in this group. |  | 0.0 (NA) — Only 1 subject was included in this group. | 20.0 (0.0) | 0.0 (NA) — Only 1 subject was included in this group. | -20.0 (NA) — Only 1 subject was included in this group. |  | 10.0 (NA) — Only 1 subject was included in this group.

12. Secondary Outcome: Change From Baseline to End of Treatment in Electrocardiogram (ECG) Parameters
Description: Change from baseline to end of treatment in ECG parameters - QRS duration, QT interval, QTcF and QTcB
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 3 | 2 | 1
ms
  QRS duration | -4.0 (8.5) | 4.0 (0.0) | 2.0 (2.3) | 2.0 (8.5) | -1.5 (3.0) | 0.7 (5.0) | -4.0 (5.7) | 0.0 (NA) — Only 1 subject was included in this group.
  QT interval | -7.0 (18.4) | 19.0 (9.9) | -5.5 (27.2) | 5.5 (27.2) | -5.0 (19.2) | -13.3 (16.2) | 7.0 (7.1) | -20.0 (NA) — Only 1 subject was included in this group.
  QTcF | -12.9 (4.4) | 12.8 (19.8) | 0.1 (24.4) | 11.0 (20.4) | -3.7 (14.5) | -10.3 (29.3) | 17.1 (4.5) | -2.9 (NA) — Only 1 subject was included in this group.
  QTcB | -16.0 (2.8) | 9.0 (25.5) | 3.5 (31.8) | 13.9 (21.4) | -2.6 (22.8) | -8.2 (37.3) | 23.0 (2.9) | 8.2 (NA) — Only 1 subject was included in this group.

13. Secondary Outcome: Change From Baseline to End of Treatment in HbA1c
Description: Change from baseline to end of treatment in HbA1c (%). LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: Data only available for 2 patients in the Placebo (adult) arm. Data only available for 3 patients in OLE I (Placebo -> Tesomet 0.125/25 mg). 5 patients started on Tesomet 0.25/25mg in OLE II however 1 subject discontinued early without any further observations and data are therefore only available from 4 subjects.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 2 | 5 | 4 | 4 | 3 | 4 | 1
Percentage of HbA1c | 0.11 (0.13) | 0.15 (0.21) | 0.06 (0.05) | 0.15 (0.24) | 0.12 (0.26) | 0.10 (0.17) | 0.00 (0.12) | 0.00 (NA) — Only 1 subject was included in this group.

14. Secondary Outcome: Change From Baseline to End of Treatment in Insulin
Description: Change from baseline to end of treatment in insulin (mIU/L). LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 2 | 5 | 4 | 4 | 3 | 4 | 1
mIU/L | 2.67 (10.93) | 1.50 (10.61) | 1.95 (13.85) | -10.32 (17.20) | 13.14 (22.15) | 4.93 (5.25) | -1.35 (24.56) | -5.90 (NA) — Only 1 subject was included in this group.

15. Secondary Outcome: Change From Baseline to End of Treatment in Fasting pl. Glucose, Triglycerides, Low-density Lipoprotein (LDL) and High-density Lipoprotein (HDL) Cholesterol
Description: Change from baseline to end of treatment in fasting pl. glucose (mmol/L), triglycerides (mmol/L), LDL and HDL cholesterol (mmol/L). LOCF.
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 2 | 5 | 4 | 4 | 3 | 4 | 1
mmol/L
  Fasting pl. glucose | 0.27 (0.59) | 0.30 (0.14) | -0.20 (0.58) | -0.30 (0.29) | 1.07 (1.19) | 0.37 (0.31) | 0.60 (0.35) | -0.40 (NA) — Only 1 subject was included in this group.
  Triglycerides | -0.07 (0.29) | -0.02 (0.06) | 0.56 (1.32) | -1.33 (1.54) | -0.54 (1.23) | 0.38 (0.14) | -0.13 (0.26) | 0.13 (NA) — Only 1 subject was included in this group.
  LDL cholesterol | -0.16 (0.44) | -0.12 (0.32) | 0.16 (0.21) | -0.32 (0.99) | -0.02 (0.43) | -0.01 (0.43) | 0.10 (0.32) | -0.25 (NA) — Only 1 subject was included in this group.
  HDL cholesterol | -0.10 (0.20) | -0.17 (0.01) | -0.03 (0.18) | -0.03 (0.17) | 0.16 (0.22) | 0.22 (0.11) | -0.05 (0.05) | -0.14 (NA) — Only 1 subject was included in this group.

16. Secondary Outcome: Number of Subjects With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Number of subjects with Adverse Events and Serious Adverse Events
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271
Measure: Count of Participants; unit: Participants
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
Number analyzed (Participants) | 6 | 3 | 5 | 4 | 4 | 4 | 5 | 1
Participants
  Subjects with at least one AE | 6 | 3 | 5 | 3 | 4 | 4 | 5 | 1
  Subjects with at least one SAE | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: DB Step 1: Day 1 to Day 91; DB Step 2: Day 1 to Day 91; OLE I: Day 91 to Day 181; OLE II: Day 181 to Day 271.
Arm/Group | Tesomet 0.50/50 mg | Placebo (Adult) | Tesomet 0.125/25 mg (DB) | Placebo (Adolescent) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg | Placebo -> Tesomet 0.125/25 mg | Tesomet 0.25/25 mg | Tesomet 0.125/25 mg (OLE II)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/5 | 0/4 | 0/4 | 0/4 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/3 | 0/5 | 0/4 | 0/4 | 0/4 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 5/5 | 3/4 | 4/4 | 4/4 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesomet 0.50/50 mg (N=6) | Placebo (Adult) (N=3) | Tesomet 0.125/25 mg (DB) (N=5) | Placebo (Adolescent) (N=4) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg (N=4) | Placebo -> Tesomet 0.125/25 mg (N=4) | Tesomet 0.25/25 mg (N=5) | Tesomet 0.125/25 mg (OLE II) (N=1)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesomet 0.50/50 mg (N=6) | Placebo (Adult) (N=3) | Tesomet 0.125/25 mg (DB) (N=5) | Placebo (Adolescent) (N=4) | Tesomet 0.125/25 mg -> Tesomet 0.125/25 mg (N=4) | Placebo -> Tesomet 0.125/25 mg (N=4) | Tesomet 0.25/25 mg (N=5) | Tesomet 0.125/25 mg (OLE II) (N=1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatillomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Negativism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03149445/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03149445/SAP_001.pdf